CLINICAL TRIAL: NCT06010407
Title: Examining the Attitudes of Physiotherapists on Patient Psychology: the Use of Psychology Methods and Psychology Education.
Brief Title: Examining the Attitudes of Physiotherapists on Patient Psychology
Status: Completed | Type: Observational
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Other Study IDs: Uskudar51
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Psychology, Social; Psychological
Keywords: physiotherapist; attitude
MeSH Terms: conditions — Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — * Working Alliance Inventory
  * Attitude Towards Psychiatry-30 Scale

SUMMARY:
To examine the psychology methods used by physiotherapists on patient psychology and to investigate their attitudes about psychology education.

DETAILED DESCRIPTION:
The answers will be collected by asking questions to the participants with an online survey. The scales and surveys to be used are as follows:

* Working Alliance Inventory (Therapeutic Alliance Scale)
* Attitude Towards Psychiatry-30 Scale
* Questionnaires prepared by the researcher.

surveys will be sent to the participants via e-mail or phone message applications.The obtained data will be analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

* Being a physiotherapist
* Having access to a computer/tablet/phone and internet
* To have accepted the voluntary consent form that requires participation in the survey study.

Exclusion Criteria:

* Those who do not meet the participation criteria
* Those who do not approve the voluntary consent form

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: active physiotherapists
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Working Alliance Inventory | 1 day
  The therapeutic alliance is an important concept that expresses the cooperation and relationship between the therapist and the patient. This alliance includes such elements as trust, mutual understanding, openness and cooperation in the therapy process. This scale can be used to identify the strengths and weaknesses of the therapeutic relationship and to evaluate the effectiveness of interventions. The total score of the BR-WAI is calculated by adding up all of the items. Reverse items, 4, 8, 12, 16, are scored inversely: (5=1) (4=2) (2=4) (1=5). A higher score represents a stronger alliance. A subscale score for Bonds is calculated by adding questions: 1, 3, 5, 7, 9, 11, 13, 15. A subscale score for Tasks and Goals is calculated by adding questions: 2, 4, 6, 8, 10, 12, 14, 16.
Attitude Towards Psychiatry-30 Scale | 1 day
  It is a scale for attitudes in psychiatry and consists of 30 items. This scale is used among medical students, physicians, nurses, and other healthcare professionals working in psychiatry. The Attitude Towards Psychiatry-30 is designed to assess attitudes about psychiatric diseases and their treatments. These attitudes cover topics such as what psychiatric illnesses are, treatment methods, and how people with psychiatric illness should be treated.Attitude Towards Psychiatry-30 is used in psychiatric healthcare in many countries.ATP-30 focuses on attitudes and views of psychiatry with 30 questions. There are 5 choices for each question: strongly agree, agree, neutral, disagree, and strongly disagree. It contains 30 Likert-scale items, 5 means strongly agree and 1 means strongly disagree.

CONTACTS AND LOCATIONS:
Overall Officials: Lobana chiah, Study Chair — Uskudar University
Locations (1):
- Uskudar university, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeVahl JM, Mulligan EP, Simpkins SD, Hynan LS. Physical Therapists' Perspectives on Lifelong Learning. J Allied Health. 2020 Fall;49(3):215-220. PMID 32877480
- [Background] da Silva TM, Costa Lda C, Garcia AN, Costa LO. What do physical therapists think about evidence-based practice? A systematic review. Man Ther. 2015 Jun;20(3):388-401. doi: 10.1016/j.math.2014.10.009. Epub 2014 Oct 24. PMID 25458142
- [Background] Lonsdale C, Hall AM, Williams GC, McDonough SM, Ntoumanis N, Murray A, Hurley DA. Communication style and exercise compliance in physiotherapy (CONNECT): a cluster randomized controlled trial to test a theory-based intervention to increase chronic low back pain patients' adherence to physiotherapists' recommendations: study rationale, design, and methods. BMC Musculoskelet Disord. 2012 Jun 15;13:104. doi: 10.1186/1471-2474-13-104. PMID 22703639
- [Background] Nicholls DA, Gibson BE. Physiotherapy as a complex assemblage of concepts, ideas and practices. Physiother Theory Pract. 2012 Aug;28(6):418-9. doi: 10.3109/09593985.2012.692557. No abstract available. PMID 22765211
- [Background] Lancelott-Redfern C, Quinlan K. A physiotherapist's life. Br Dent J. 2014 Jun 13;216(11):610-1. doi: 10.1038/sj.bdj.2014.464. No abstract available. PMID 24923923